CLINICAL TRIAL: NCT02982512
Title: Effects of Different Concentrations of Dexmedetomidine on Basal Ganglia Neuronal Activity (Local Field Potentials) in Parkinson's Disease
Brief Title: Dexmedetomidine on Basal Ganglia Neuronal Activity in Parkinson's Disease
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: DEXPAR
Record Dates: First submitted 2016-11-28; First posted 2016-12-05 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Dexmedetomidine; Deep Brain Stimulation; Parkinson Disease
Keywords: Potential local fields; Subthalamic neuronal activity
MeSH Terms: conditions — Parkinson Disease | interventions — Dexmedetomidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control recording (No Intervention): Recording of local field potentials without drugs from the deep brain stimulator
- Dexmedetomodine recording (Experimental): Recording of local field potentials at different dexmedetomidine concentrations from the deep brain stimulator
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — Administration of dexmedetomidine a different concetrations
  Other Names: Dexdor
  Arms: Dexmedetomodine recording

SUMMARY:
The implantation of a deep brain stimulator (DBS) is an established option to improve the symptoms of Parkinson's disease (PD) in patients that do not respond adequately to medical therapy. Most centers perform this surgery using a technique that involves microelectrode recording (MER) of neuronal activity for localization of the target nucleus, microstimulation of identified targets, and neurological intraoperative testing in a cooperative patient.

Dexmedetomidine, a α2-adrenergic receptors agonist, is a potent anxiolytic that acts at subcortical areas of the brain without involving GABA receptors. It provides excellent sedation without respiratory depression; also, it has an analgesic component and a predictable hemodynamic response. Low maintenance doses do not appear to interfere with MER. The possible effect of dexmedetomidine in the PD symptoms is still unclear.

DETAILED DESCRIPTION:
The implantation of a deep brain stimulator (DBS) is an established option to improve the symptoms of Parkinson's disease (PD) in patients that do not respond adequately to medical therapy. Most centers perform this surgery using a technique that involves microelectrode recording (MER) of neuronal activity for localization of the target nucleus, microstimulation of identified targets, and neurological intraoperative testing in a cooperative patient. This surgery is usually performed in two stages. In the first stage, and under conscious sedation (CS), the target nucleus is localized and the DBS is implanted. About 5 days later, and under general anaesthesia, a programmable pulse generator is implanted and connected to the DBS.

The anesthetic approach varies depending on the institution, ranging from local anesthesia only with monitored care, conscious sedation, and the "asleep-awake" or "asleep-awake-asleep" technique. But sedative drugs can affect the quality of MER by suppressing the firing rate of basal ganglia structures, and alter PD symptoms. Propofol is the drug most commonly used. Its real influence on the quality of MER and PD symptoms is still today controversial. In recent years, some studies have suggested using dexmedetomidine as the main sedative agent for this intervention. Dexmedetomidine, a α2-adrenergic receptors agonist, is a potent anxiolytic that acts at subcortical areas of the brain without involving GABA receptors. It provides excellent sedation without respiratory depression; also, it has an analgesic component and a predictable hemodynamic response. Low maintenance doses do not appear to interfere with MER. The possible effect of dexmedetomidine in the PD symptoms is still unclear. All these characteristics make it a good choice for sedation of PD patients undergoing DBS surgery.

Studying the influence of anesthetic drugs on basal ganglia activity and PD motor symptoms in humans and in a clinical setting is complicated. First, it is difficult to establish a control group to compare effects in different nuclei. There is some data concerning clinical outcomes (clinical symptoms or long term stimulation parameters) but without electrophysiological data. MERs data has been compared between different patients or in the same patient but between contralateral targets. Few studies analyze electrophysiological data with or without one sedative drug in the same target.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing placement of DBS for PD in two phases.
* The patient must be of legal age (> 17 years old).
* The patient or his representative has consented to participate in the study.
* The patient should, in the investigator's opinion, be able to cooperate during the procedure.

Exclusion Criteria:

* Known liver disease.
* Pregnant or nursing women.
* History of hypersensitivity to dexmedetomidine.
* Heart block (2nd or 3rd degree), without pacemaker.
* Symptomatic hypotension.
* Severe stroke or other neurological deficits that may impair adequate cooperation or observation of the study endpoints.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-09 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Beta activity (15-35 Hz) | Control and dexmedetomidine exposure (around 300 min of continuous recording)
  Global power in the beta band (15-35 Hz) of the electrical oscillatory activity from deep brain structures.

SECONDARY OUTCOMES:
Bispectral index scales (a single dimensionless number ranges from 0 - 100) | Control and dexmedetomidine exposure (around 300 min of continuous recording)
  Weighted sum of several electroencephalographic subparameters, including a time domain, frequency domain, and high order spectral subparameters

CONTACTS AND LOCATIONS:
Overall Officials: Martinez-Simon Antonio, MD, PhD, Principal Investigator — Staff of Anesthesiology Department
Locations (1):
- Clínica Universidad de Navarra, Pamplona, Navarre, Spain